CLINICAL TRIAL: NCT04325633
Title: Efficacy of Addition of Naproxen in the Treatment of Critically Ill Patients Hospitalized for COVID-19 Infection
Acronym: ENACOVID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stop inclusions for insufficient recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200387
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Naproxen; Nonsteroidal anti-inflamatory drug
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: Naproxen (Experimental): Administration of naproxen 250 mg twice and lansoprazole 30 mg daily for prevention of gastropathy induced by stress or a nonsteroidal anti-inflammatory drug (NSAID) in addition to standard of care (SOC)
  Interventions: Drug: 1: Naproxen; Drug: 2: Standard of care
- 2: Standard of care (Placebo Comparator): Standard of care
  Interventions: Drug: 2: Standard of care

INTERVENTIONS:
Drug: 1: Naproxen — Description : Administration of naproxen 250 mg twice and lansoprazole 30 mg daily for prevention of gastropathy induced by stress or a nonsteroidal anti-inflammatory drug (NSAID) in addition to standard of care (SOC)
  Arms: 1: Naproxen
Drug: 2: Standard of care — Standard of care

SUMMARY:
The symptoms of respiratory distress caused by COVID-19 may be reduced by drugs combining anti-inflammatory and antiviral effects. This dual effect may simultaneously protect severely-ill patients and reduce the viral load, therefore limiting virus dissemination We want to demonstrate the superiority of naproxen (anti-inflamatory drug) treatment addition to standard of care compared to standard of care in term of 30-day mortality.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is due to SARS-CoV-2 infection. (1,2) The exacerbated inflammatory response in COVID-19 infected critically ill patients calls for appropriate anti inflammatory therapeutics combined with antiviral effects. Thus, drugs combining anti-inflammatory and antiviral effects may reduce the symptoms of respiratory distress caused by COVID-19. This dual effect may simultaneously protect severely ill patients and reduce the viral load, therefore limiting virus dissemination. Naproxen, an approved anti-inflammatory drug, is an inhibitor of both cyclo oxygenase (COX-2) and of Influenza A virus nucleoprotein (NP). The NP of Coronavirus (CoV), positive-sense single-stranded viruses, share with negative-sense single-stranded viruses as Influenza the ability to bind to- and protect genomic RNA by forming self-associated oligomers in a helical structure with RNA. Naproxen was shown to bind the Influenza A virus NP making electrostatic and hydrophobic interactions with conserved residues of the RNA binding groove and C terminal domain. (3) Consequently, naproxen binding competed with NP association with viral RNA and impeded the NP self-association process which strongly reduced viral transcription/replication. This drug may have the potential to present antiviral properties against SARS-CoV-2 suggested by modelling work based on the structures of CoV NP. The high sequence conservation within the coronavirus family, including severe acute respiratory syndrome (SARS-CoV) and the present SARSCoV-2 coronavirus allows to perform this comparison. (4) A recent clinical trial shown that the combination of clarithromycin, naproxen and oseltamivir reduced mortality of patients hospitalized for H3N2 Influenza infection. (5). Inappropriate inflammatory response in CODIV-19 patients was demonstrated in a recent study where Intensive Care Unit (ICU) patients had higher plasma levels of IL2, IL7, IL10, GSCF, IP10, MCP1, MIP1A, and TNF? compared with non-ICU patients.(2) We suggest that naproxen could combine a broad-spectrum antiviral activity with its well-known anti inflammatory action that could help reducing severe respiratory mortality associated with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infected patient
* Age 18 years or older
* Presence of pneumonia
* PaO2/FiO2 < 300 mm Hg or SpO2 < 93% in air ambient or need to supplementary oxygen administration in order to maintain SpO2 range in [94-98%] or lung infiltrates > 50%
* Medical insurance

Exclusion Criteria:

* Presence of do-not-resuscitate order
* Pregnancy
* Prisoners
* Known Naproxen allergy or intolerance
* Severe renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Mortality all causes at day30 | at day30

SECONDARY OUTCOMES:
Number of days alive free of mechanical ventilation | during 30 days after randomization
Number of days alive outside | during 30 days after randomization
Number of days alive outside hospital | during 30 days after randomization
Maximal changes in Sofa score | in the first 7 days after randomization
Time to negativation of virus titer in the nasopharyngeal aspirate (NPA) | during 90 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ADNET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Réanimation médico-chirurgicale, Avicenne Hospital, Bobigny
  - Urgences, Avicenne Hospital, Bobigny